CLINICAL TRIAL: NCT00784472
Title: Visceral Pain Originating From the Upper Urinary Tract - a Randomized Controlled Trial on the Effect of Morphine and Oxycodone in Patients Undergoing Percutaneous Nephrolithotomy (PCNL)
Brief Title: Visceral Pain From the Upper Urinary Tract - a Trial on the Effect of Morphine and Oxycodone in Patients Undergoing PCNL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Katja venborg Pedersen (Other)
Collaborators: Aalborg University Hospital (Other)
Responsible Party: Sponsor-Investigator, Katja venborg Pedersen, MD, Fredericia Hosptial
Organization: Fredericia Hosptial (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VEN 1
Record Dates: First submitted 2008-10-27; First posted 2008-11-04 (Estimated); Last update posted 2012-07-09 (Estimated); Status verified 2012-07

CONDITIONS: Kidney Stones
Keywords: PCNL; oxycodone; morphine; visceral pain
MeSH Terms: conditions — Kidney Calculi; Visceral Pain | interventions — Oxycodone; Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- oxycodone (Active Comparator)
  Interventions: Drug: oxycodone
- morphine (Active Comparator)
  Interventions: Drug: morphine

INTERVENTIONS:
Drug: oxycodone — intravenous according to patients weight, pn.
  Other Names: oxynorm N02A A05
  Arms: oxycodone
Drug: morphine — intravenous administration according to patients weight, pn.
  Other Names: morphine SAD N02 AA 01
  Arms: morphine

SUMMARY:
The purpose of this study is to investigate the effect of oxynorm versus morphine after operation for kidney stone (PCNL). In addition the relationship between pain symptoms and referred sensory and trophic changes will be examined in the patients before and after the operation.Finally a blood sample is analysed to investigate pharmaca-genetics.

DETAILED DESCRIPTION:
Primary outcome: the amount of opioid (morphine or oxynorm) used the first 4 hours postoperatively.

Secondary outcome: side effect to the opioids, pain score, pain threshold to electrical stimulation and pressure before and after operation, pharmacogenetics, size of referred pain area.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* Indication for PCNL

Exclusion Criteria:

* Malignant disease in the upper urinary tract
* Allergy to morphine or oxycodone
* Use of opioids the last 48 hours before PCNL
* Pregnancy
* Nursing mothers
* Present JJ-stent in the ureter
* Previous urinary stone disease on the opposite site

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2008-12; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Amount of analgetics used | four hours postoperatively

SECONDARY OUTCOMES:
Side effects | four hours postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Palle Osther, Professor, Study Chair — Hospital Little Belt, Fredericia; katja Venborg Pedersen, MD, Principal Investigator — Hospital Little Belt, Fredericia
Locations (1):
- Hospital Little Belt, Fredericia, Fredericia, Denmark